CLINICAL TRIAL: NCT05593614
Title: A Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled, Phase 2 Study to Assess the Efficacy and Safety of ATX01 (Topical Amitriptyline Hydrochloride 10% and 15% w/w) in Comparison to Placebo, in Cancer Survivor Adult Patients With Chemotherapy-induced Peripheral Neuropathy (CIPN)
Brief Title: Efficacy and Safety of ATX01 in Adult Patients With CIPN (Chemotherapy-induced Peripheral Neuropathy)
Acronym: ACT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AlgoTherapeutix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATX01-22-01-CIPN; 2022-000435-23 (EudraCT Number)
Record Dates: First submitted 2022-10-21; First posted 2022-10-25 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-01

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ATX01 10% (Experimental): A bottle of hydrogel formulation containing 10% amitriptyline hydrochloride w/w for topical use on the hands and/or feet, morning and night for 3 months.
  Interventions: Drug: ATX01 10%
- ATX01 15% (Experimental): A bottle of hydrogel formulation containing 15% amitriptyline hydrochloride w/w for topical use on the hands and/or feet, morning and night for 3 months.
  Interventions: Drug: ATX01 15%
- ATX01 Placebo (Placebo Comparator): A bottle of hydrogel formulation containing no active ingredient, for topical use on the hands and/or feet, morning and night for 3 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ATX01 10% — A 100 mL bottle of hydrogel formulation containing 10% amitriptyline hydrochloride w/w
  Arms: ATX01 10%
Drug: ATX01 15% — A 100 mL bottle of hydrogel formulation containing 15% amitriptyline hydrochloride w/w
  Arms: ATX01 15%
Drug: Placebo — A 100 mL bottle of hydrogel formulation containing no active substance
  Arms: ATX01 Placebo

SUMMARY:
The purpose of this clinical trial is to compare the efficacy of twice daily applications of ATX01 (10% & 15%) versus placebo during a 12-week treatment period in treating chemotherapy-induced peripheral neuropathy (CIPN) in adult cancer survivor patients.

ELIGIBILITY:
Inclusion criteria

1. Male or female patients of 18 years and older.
2. Patients having signed a written informed consent prior to any study-related procedure.
3. Body mass index of 18 to 35 kg/m2 (inclusive).
4. With an estimated life expectancy ≥6 months at study entry.
5. Patients with painful sensory CIPN resulting from prior treatment of cancer with taxanes or platins. A diagnosis of CIPN should be supported by i) onset of pain in hands or feet after exposure to taxanes or platins, ii) presence of painful symptoms in a symmetrical stocking and/or glove distribution, AND iii) painful symptoms may be accompanied by nonpainful symptoms (eg, tingling/pins and needles intensity and numbness intensity).
6. Patients who have stopped their chemotherapy treatment with taxanes or platins or any other neurotoxic chemotherapy for ≥24 weeks at the time of the screening visit.
7. Patients with CIPN pain for ≥24 weeks at the time of the screening visit.
8. Patients with a mean value of pain intensity ≥4 and ≤9 in target study extremities (left and right feet or left and right hands) on the 11 point NPRS at baseline. Non target extremities can be treated regardless of the pain intensity.
9. Patients with symmetrical stocking or glove distribution pain, NPRS (≤1 point difference) in the target study extremities at screening.
10. Neuropathic Pain (DN4) score ≥4 in the target study extremities (hands or feet) at the screening visit
11. Treatment naïve patients or patients in whom any prior CIPN treatment (except oral amitriptyline [AMT]) has not been modified during the 4 weeks preceding the screening visit and is planned to be maintained at the same regimen during the course of the study (prior treatment includes pharmacological and nonpharmacological treatments).
12. Male patients should agree to use a condom along with another medically acceptable contraceptive method, where applicable according to local guidelines, if he is engaged in sexual activity with a woman of childbearing potential (WOCBP) from the day of the signature of the informed consent and up to 90 days after the End-of-Study (EoS) Visit. Male patients should agree not to donate sperm until 30 calendar days after the last dose of study drug.
13. Females must comply with the following in order to be enrolled:

    1. WOCBP with negative serum pregnancy test results can be enrolled only if willing to use an acceptable contraceptive method, ie, oral contraceptives, patch contraceptives, injection contraceptives, implantable hormonal contraceptives, male condom with intravaginal spermicide, diaphragm or cervical cap with spermicide, vaginal contraceptive ring, intrauterine device or system, surgical sterilization (hysterectomy, bilateral oophorectomy, and/or bilateral salpingectomy), tubal ligation/occlusion, vasectomized partner, or sexual abstinence, if this is the patient's current practice, from at least 14 days prior to the screening visit and throughout the study and for at least 30 days after the completion of the study.
    2. Or surgically sterilized for at least 6 months.
    3. Or menopausal for at least 1 year.

Exclusion criteria

1. Patients who are not compliant in completion of pain ratings during the screening period. Patients having <5 of 7 records of average pain intensity in the target study extremities from Day -7 to Day -1 will be excluded. If a patient misses records of 2 days out of 7 days, the patient will be included in the study; however, patients missing 3 or more days of records will be excluded from the study.
2. Clinical evidence of a preexisting painful peripheral neuropathy resulting from another cause than chemotherapy, eg, diabetic neuropathy, posttraumatic neuropathy, carpal/tarsal tunnel syndrome, radiculopathy, spinal stenosis, brachial plexopathy, or other preexisting symptomatic neuropathy due to alcoholism, vitamin B deficiency, hypothyroidism, human immunodeficiency virus. Patients may be included in the study, providing that pain appeared after chemotherapy, while other non-painful symptoms could have been present before start of chemotherapy.
3. Skin irritation, or lesions (eg open skin wounds, infections, inflammations, or exfoliative dermatitis) of any type on the hands or feet (or only on the hands if the study drug is not applied on the feet and vice versa [only on the feet if the study drug is not applied on the hands]).
4. Presence of glaucoma.
5. Presence of urinary retention (or significant prostatic hypertrophy at risk of urinary retention).
6. Angina or myocardial infarction in the year preceding screening visit.
7. History and/or presence of major depressive episode. Patients with a medical history of bipolar disorder, alcohol abuse, or psychotic disorder are also excluded.
8. Patients who are at significant risk of suicide, or are a danger to self or others, in the opinion of the investigator, based upon clinical interview and the C-SSRS at screening and baseline. Affirmative answer to suicidal ideation questions 4 or 5 within the last 6 months and / or suicidal behavior (actual attempt, interrupted attempt, aborted attempt, and/or preparatory acts/behavior) within the last 2 years are exclusionary.
9. Pregnant or lactating women.
10. Abnormality in the 12-lead electrocardiogram (ECG) at screening that in the opinion of the investigator increases the risk of participating in the study, such as a corrected QT Fridericia (QTcF) interval >430 msec for males or >450 msec for females.
11. A history of additional risk factors for Torsade de Pointe (eg, heart failure, hypokalemia, family history of long QT syndrome).
12. The use of concomitant medications within 24 weeks prior to Day 1 and/or during the study or the equivalent of 5 half-lives that prolong the QT/QTc interval, eg, Class 1 antiarrhythmics (eg, quinidine, disopyramide, procainamide) and Class 3 antiarrhythmics (eg, amiodarone, sotalol), first generation antihistamines (such as diphenhydramine, hydroxyzine, astemizole, terfenadine, and ebastine), antipsychotics known to prolong QT interval, and antimalarials (eg, mefloquine, quinine), tricyclic antidepressants (eg, AMT), tetracyclic antidepressants (eg, maprotiline), cisapride.
13. The use of monoamine oxidase inhibitors within 24 weeks (or the equivalent of 5 half-lives) prior to Day 1 and/or during the study.
14. The use of opioids within 4 weeks (or the equivalent of 5 half lives) prior to Day 1 and/or during the study.
15. History of illicit drug use or confirmed drugs of abuse at screening. Positive urine drug screen for prescribed medication is allowed at the discretion of the investigator.
16. Patients likely to require neurotoxic chemotherapy treatment or any other treatment during the study, which may interfere with compliance to the protocol, ability to complete the study and study assessments except treatments authorized in inclusion criterion #11.
17. Failure to respond to more than 2 analgesics (regardless of the route of administration) from different drug classes (including antidepressants and anticonvulsants) due to lack of efficacy to treat CIPN at any time in the past. The definition of failure to respond is left to the investigator's judgement and should be understood as exclusion of patients who are non-responding to more than 2 analgesics thought to be effective for neuropathic pain that were used at therapeutic doses in the 6 months prior to screening visit.
18. Treatment with oral or topical AMT or nortriptyline in the past 4 weeks prior to baseline visit.
19. Any known hypersensitivity to AMT (regardless of the route of administration) in any salt form or to any constituent of the topical formulation.
20. Any contraindication to the use of acetaminophen/paracetamol.
21. Use of glutathione, vitamin E, or minocycline within 12 weeks of screening.
22. Any topical treatment on treated extremities for any indication, other than cosmetic use of creams and lotions, within the previous 12 weeks prior to Baseline visit.
23. Any topical treatment for pain on extremities including use of:

    1. over-the-counter capsaicin on extremities within 2 weeks of Baseline visit,
    2. and/or Qutenza within 12 weeks of Baseline visit,
    3. and/or nonsteroidal anti-inflammatory drugs, menthol, methyl salicylate, local anesthetics within 1 week of screening.
24. Poor metabolizer for cytochrome P450 CYP2D6.
25. Intake in the 4 weeks preceding the screening visit of any strong inhibitor of cytochrome P450 CYP2D6.
26. Treatment with an investigational drug in the previous 4 weeks or greater prior to Baseline visit, according to local requirements.
27. Any condition that the investigator feels would place the patient at increased risk if the investigational therapy is initiated, such as, but not limited to, hyperthyroidism, convulsive disorder, advanced hepatic disease, pylorus, stenosis, or paralytic ileus.
28. The investigator considers the patient unfit for the study as a result of the medical interview, physical examination, or screening investigations, in particular any status or disease making the patient unable to follow instructions.
29. The patient is unable to apply the study drug on hands or feet.
30. The patient is an employee of the investigator, study site, sponsor, or CRO with direct involvement in the proposed study or other studies under the direction of the investigator, study site, or sponsor, or a family member of the site employee or the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to Week 12 in the weekly mean of the daily NPRS score assessing average pain intensity in target study extremities related to CIPN in the past 24 hours. | 12 weeks

SECONDARY OUTCOMES:
Percentage of patients achieving ≥30% pain reduction from baseline in the weekly mean NPRS average pain intensity related to CIPN at Week 12 | 12 weeks
Percentage of patients achieving ≥50% pain reduction from baseline in the weekly mean NPRS average pain intensity related to CIPN at Week 12. | 12 weeks
Mean change from baseline to each visit in tingling/pins and needles intensity and numbness intensity in target study extremities as measured by the numerical rating scale (NRS) assessing each symptom | 4 weeks, 8 weeks, 12 weeks
Proportion of patients achieving various percentages of reduction in average pain intensity in target study extremities (cumulative responder curve) throughout the study. | 4 weeks, 8 weeks, 12 weeks
Proportion of patients achieving various percentages of reduction in worst pain intensity in target study extremities (cumulative responder curve) throughout the study. | 4 weeks, 8 weeks, 12 weeks
Change from baseline to Week 4 and 8 in the weekly mean of the daily NPRS score assessing average pain intensity in target study extremities related to CIPN in the past 24 hours | 4 weeks, 8 weeks
Change from baseline to each visit in the weekly mean of the daily NPRS assessing worst pain intensity in target study extremities related to CIPN in the past 24 hours | 4 weeks, 8 weeks, 12 weeks
Percentage of patients with at least "improved" on the Patient Global Impression of Change (PGI-C) at each visit | 4 weeks, 8 weeks, 12 weeks
Mean change from baseline to each visit in pain interference with daily life using the Brief Pain Inventory Short Form questionnaire (BPI-SF item 9 only) | 4 weeks, 8 weeks, 12 weeks
Mean change from baseline to each visit in the calculated mean NPRS average pain intensity in the nontarget study extremities | 4 weeks, 8 weeks, 12 weeks
Mean change from baseline to Week 12 in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-CIPN 20-item scale (EORTC QLQ CIPN20) | 12 weeks
Use of rescue medication including the proportion of patients using rescue medication, the frequency, and amount used | Up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (43):
- United States (8):
  - South Lake Pain Institute, Clermont, Florida
  - MGM Medical Care Research & Rehab, LLC, Miami, Florida
  - Medsol Clinical Research Center, Inc, Port Charlotte, Florida
  - Knight Neurology - Clinical Research, Rockledge, Florida
  - Neuroscience Research Center, LLC., Overland Park, Kansas
  - The Center for Cancer and Blood Disorders (CCBD), Bethesda, Maryland
  - University of Rochester Medical Center, Rochester, New York
  - HD Research, Bellaire, Texas
- Belgium (5):
  - OLV Hospital Aalst: gastro-enterologie, Aalst
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent (UZ Gent), Ghent
  - UZ Leuven / Campus Pellenberg / Pain Center, Pellenberg
  - CHU UCL Namur - site Godinne, Yvoir
- Czechia (3):
  - Clinitrial s.r.o., Prague
  - Praglandia s.r.o., Prague
  - Nemocnice Teplice, Teplice
- France (8):
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Institute Bergonie, Bordeaux
  - CHU de Montpellier, Hôpital Saint Eloi, Montpellier
  - Groupe Hospitalier Paris Saint Joseph, Paris
  - CHU POITIERS, Hépato-Gastro Entérologie, Poitiers
  - GODINOT Institute, Reims
  - Strasbourg Oncologie Liberale, Strasbourg
  - Hôpital Foch, Suresnes
- Italy (6):
  - Gemelli Molise S.p.a., Campobasso
  - Istituto Scientifico Romagnolo per lo Studio e La cura dei Tumori Srl (IRST), Meldola
  - Fondazione IRCCS Ca' Granda Ospedale -. Maggiore Policlinico, Milan
  - ASST Monza - Ospedale S. Gerardo di Monza, Monza
  - Fondazione IRCCS Policlinico San Matteo - Universita degli Studi di Pavia, Pavia
  - Azienda Ospedaliera San Camillo-Forlanini, Roma
- Poland (4):
  - Przychodnia Lekarska "Komed" Roman Karaszewski Oddzial Chemioterapii Jednego Dnia, Konin
  - Instytut "Centrum Zdrowia Matki Polki" Klinika Onkologii, Lodz
  - Niepubliczny Zaklad Opieki Zdrowotnej Poradnia Leczenia Bolu Przewleklego, Tychy
  - ClinHouse sp z o.o. - ClinHouse Centrum Medyczne, Zabrze
- Spain (9):
  - Hospital de la Santa Creu I de Sant Pau, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Complejo Hospitalarion de Jaen, Jaén
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Ruber Internacional, Madrid
  - Madrid Sanchinarro Hospital, Madrid
  - Hospital Universitari Sant Joan de Reus, Reus
  - Unidad de Investigacion Clinica FINCIVO, Valencia